CLINICAL TRIAL: NCT02144259
Title: The Impact of Contraception on Postpartum Weight Loss: a Prospective Study
Brief Title: The Impact of Contraception on Postpartum Weight Loss
Acronym: PPWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 813000
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Weight
MeSH Terms: conditions — Body Weight | interventions — Medroxyprogesterone Acetate; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DMPA group (Active Comparator): Subjects randomized to receive DepoProvera(DMPA) immediately post-partum.
  Interventions: Drug: DMPA immediately postpartum
- Implanon group (Active Comparator): Subjects randomized to receive Implanon immediately post-partum.
  Interventions: Drug: Implanon immediately postpartum
- Control group (No Intervention): Subjects selecting their own method of contraception or no contraception.

INTERVENTIONS:
Drug: DMPA immediately postpartum — DMPA is an intramuscular injection of 150mg of depot medroxyprogesterone acetate.
  Other Names: DepoProvera, depot medroxyprogesterone acetate (DMPA)
  Arms: DMPA group
Drug: Implanon immediately postpartum — Implanon ® is a subdermal implant that contains 68mg of etonogestrel.
  Other Names: etonogestrel implant
  Arms: Implanon group

SUMMARY:
This is a prospective mixed methods study to assess weight changes in women randomized to receive Implanon ® or Depo Provera® (DMPA) immediately postpartum compared to women who choose non-hormonal contraception or no contraception immediately postpartum. After enrollment, subjects return for a visit at 3, 6 and 12 months postpartum to be asked a series of questions, take a pregnancy test, and be weighed. Total length of participation for each subject is 1 year or until pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Aged 18-45 at enrollment (inclusive)
* Immediately postpartum of a live singleton infant, 37 weeks gestation, at HUP
* Desiring to delay another pregnancy for 6 months
* Willing and able to follow the study protocol

Exclusion Criteria:

* Breastfeeding during study participation
* Plans for relocation outside of Philadelphia in the next six months
* Plans for use of weight loss medication or diet pills in the next six months
* Women who wish to start Implanon ® or DMPA prior to discharge but who do not want to be randomized. 5. Issues or concerns in the judgment of the investigator that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney A Schreiber, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DMPA Group | Implanon Group | Control Group
Started | 33 | 33 | 34
Completed | 23 | 28 | 16
Not Completed | 10 | 5 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMPA Group | Implanon Group | Control Group | Total
Number analyzed (Participants) | 33 | 33 | 34 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.06 (4.68) | 22.42 (3.81) | 26.59 (5.42) | 24.02 (4.63)
Gender [Count of Participants; unit: Participants]
  Female | 33 | 33 | 34 | 100
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 34 | 100

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Weight will be measured at 6 months postpartum. Percent weight change will be compared amongst the groups
Time Frame: 6 months from postpartum (baseline)
Measure: Mean (Standard Deviation); unit: percent weight lost
Arm/Group | DMPA Group | Implanon Group | Control Group
Number analyzed (Participants) | 23 | 28 | 16
percent weight lost | 3.2 (9.1) | 6.8 (8.1) | 7.0 (10.2)
Statistical Analysis 1: Comparison: DMPA Group vs Implanon Group vs Control Group; Because the expected amount of postpartum weight loss in non-breastfeeding women is not documented in the literature, we chose a sample size that would enable us to detect a one standard deviation difference in weight loss between the 3 groups at the primary 6 month endpoint. We used generalized estimating equations (GEEs) to test differences among all 3 groups over all the study periods; Test type: Superiority or Other; p < 0.05, GEE

2. Secondary Outcome: Pregnancy Rate
Description: The secondary outcome variable is pregnancy rate. Pregnancy testing will occur at 3, 6 and 12 months postpartum or at any time that a participant felt that she might be pregnant.
Time Frame: 1 year
Measure: Number; unit: number of pregnancies
Arm/Group | DMPA Group | Implanon Group | Control Group
Number analyzed (Participants) | 23 | 28 | 16
number of pregnancies | 1 | 1 | 4

3. Other Pre Specified Outcome: Contraceptive Satisfaction
Description: Satisfaction will be measured in response to the question, "How satisfied are you with your current birth control method?" This question will be asked to the participant at the 6 month follow-up visit. Answer choices that participants could choose from range from "Very Good" to "Very Poor". "Good" or "Very Good" responses will be analyzed as having been satisfied with the method.
Time Frame: 1 year
Measure: Number; unit: percentage of women satisfied w. method
Arm/Group | DMPA Group | Implanon Group | Control Group
Number analyzed (Participants) | 23 | 28 | 16
percentage of women satisfied w. method | 74 | 89 | 75
Statistical Analysis 1: Comparison: DMPA Group vs Implanon Group vs Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | DMPA Group | Implanon Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/34

LIMITATIONS AND CAVEATS:
First, we chose to exclude nursing women. Second, we had a small sample with power to detect one standard deviation difference in weight loss. Third, all data were collected prospectively,thus we did not have each participant's pre-pregnancy weight.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No